CLINICAL TRIAL: NCT03479801
Title: Comparative Study of Surgical Results in Endoscopic Thyroidectomy Via Oral Approach, Via Breast Approach and Conventional Open Thyroidectomy
Brief Title: Comparative Study in Oral, Breast Approach and Open Thyroidectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 87783760
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-02

CONDITIONS: Thyroid Neoplasms
MeSH Terms: conditions — Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Conventional Open: Conventional open thyroidectomy group (thyroid neoplasms patients who underwent conventional thyroidectomy procedure with or without postoperative central node dissection)
  Interventions: Procedure: Thyroid Surgical Methods
- Transoral Endoscopic Surgery: Transoral endoscopic thyroidectomy via vestibular approach group (thyroid neoplasms patients who underwent conventional thyroidectomy procedure with or without postoperative central node dissection)
  Interventions: Procedure: Thyroid Surgical Methods
- Endoscopic Thyroidectomy via Breast: Endoscopic thyroidectomy via breast approach or bilateral areola approach group (thyroid neoplasms patients who underwent conventional thyroidectomy procedure with or without postoperative central node dissection)
  Interventions: Procedure: Thyroid Surgical Methods

INTERVENTIONS:
Procedure: Thyroid Surgical Methods — Different methods of thyroid surgery, including conventional open thyroidectomy, transoral endoscopic thyroidectomy via vestibular approach, and endoscopic thyroidectomy via breast approach.

SUMMARY:
Purpose: Total endoscopic thyroidectomy including oral approach and breast approach has excellent cosmetic and several functional results. Many patients, especially women, undergoing thyroid surgery are concerned about the postoperative cosmetic appearance of the neck. The procedure of total endoscopic thyroidectomy by breast approach only left three incisions, while by oral approach did not leave any incisions in the body surface, which is scarless in the neck, involved with a higher cosmetic result. However, the long-term property evaluation of total endoscopic thyroidectomy was not confirmed. The purpose of our study was to evaluate the surgical results of total endoscopic thyroidectomy (transoral approach and breast approach) versus conventional open thyroidectomy.

DETAILED DESCRIPTION:
Purpose: Total endoscopic thyroidectomy including oral approach and breast approach has excellent cosmetic and several functional results. Many patients, especially women, undergoing thyroid surgery are concerned about the postoperative cosmetic appearance of the neck. Transoral endoscopic thyroidectomy via vestibular approach (TOETVA) and endoscopic thyroidectomy via breast approach were routinely performed in our institute. The procedures of total endoscopic thyroidectomy by breast approach only left three incisions, while by oral approach did not leave any incisions in the body surface, which is scarless in the neck, involved with a higher cosmetic result. However, the comprehensive comparison between transoral approach, breast approach and conventional open method was not confirmed. The purpose of our study was to evaluate the surgical results of total endoscopic thyroidectomy (transoral approach and breast approach) versus conventional open thyroidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 15~55 years old;
2. Type: Differentiated thyroid carcinoma, diameter ≤ 2cm, cN0 or cN1a, M0;
3. Thyroid lobe was less than the second degree enlargement;
4. Thyroid benign goiter, and the diameter ≤ 6cm

Exclusion Criteria:

1. Combine the surgical history of mandibular, oral, facial, or neck;
2. It was shown by preoperative radiological examination that the thyroid cancer has local invasion, N1b, or distant metastasis.
3. Thyroid lobe was more than the third degree enlargement
4. Any medical history that probably interfere the test results or increase the disease risks
5. The patient's compliance is not very well, and cannot work as the doctors asked

Ages: 15 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Choosing to participate in a study is an important personal decision. Talk with your doctor and family members or friends about deciding to join a study. To learn more about this study, you or your doctor may contact the study research staff using the contacts about the eligibility criteria. Patients will be introduced the general information of different surgical methods, and the clinical studies.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life assessment postoperatively | 12 months after the surgery of thyroidectomy
  Physicians Global Assessment to measure quality of life was performed, and the assessment form had been verified.

SECONDARY OUTCOMES:
Cosmetic results of thyroidectomy postoperatively | 12 months after the surgery of thyroidectomy
  Visual Analog Score (1-10) for the cosmetic results (evaluated by patients) was been performed.
Surgical Complications of thyroidectomy postoperatively | 12 months after the surgery of thyroidectomy
  The rates (percentage) of surgical complications (transient or permanent Recurrent Laryngeal Nerve paralysis, transient or permanent hypoparathyroidism, Postoperative hemorrhage)
Surgical Completeness of thyroidectomy postoperatively | 12 months after the surgery of thyroidectomy
  The rates (percentage) of surgical completeness (whether or not any thyroid associated tissues left by the examination of ultrasound and Iodine-131)

CONTACTS AND LOCATIONS:
Overall Officials: Jianan Wang, MD., Study Director — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- SAHZhejiangU, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
Participants who had studied endoscopic thyroid surgeries in our department would be introduced.

REFERENCES:
- [Result] Wang Y, Yu X, Wang P, Miao C, Xie Q, Yan H, Zhao Q, Zhang M, Xiang C. Implementation of Intraoperative Neuromonitoring for Transoral Endoscopic Thyroid Surgery: A Preliminary Report. J Laparoendosc Adv Surg Tech A. 2016 Dec;26(12):965-971. doi: 10.1089/lap.2016.0291. Epub 2016 Sep 1. PMID 27585396
- [Derived] Zhu R, Yue N, Hong Y, Ye Q, Han Z, Luo Z, Xie C, Yan H, Yu X. Ectopic parathyroid adenomas in primary hyperparathyroidism: anatomical classifications, localization strategies, and case series. Int J Surg. 2026 Jan 12. doi: 10.1097/JS9.0000000000004578. Online ahead of print. PMID 41417934
- See also: The links of reference which is related with this study — http://online.liebertpub.com/doi/10.1089/lap.2016.0291